CLINICAL TRIAL: NCT03296826
Title: Prospective Cohort Study of Germline Variant Carriers With BRCA1 or BRCA2
Status: Recruiting | Type: Observational
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Okayama University (Other); Japanese Gynecologic Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: JGOG3024; UMIN000028740 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: BRCA1 and/or BRCA2 Variant Carriers; Ovarian Carcinoma; Fallopian Tube Carcinoma; Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (all subjects) for Germ-line DNA sequencing, Biospy samples(when subjects have RRSO within follow-up duration)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BRCA1/2 variant carriers: Japanese women who carry BRCA 1/2 variants.

SUMMARY:
To determine the incidence and risk factors in the development of ovarian, fallopian tube, and peritoneal cancers in Japanese women carrying Breast Cancer Susceptibility Gene (BRCA)1/2 variants.

DETAILED DESCRIPTION:
1. To estimate the incidence of ovarian, fallopian tube and peritoneal cancers in women carrying BRCA1/2 variants.
2. To investigate risk factors concerning the development of ovarian, fallopian tube, and peritoneal cancers (loci of BRCA1/2 genetic variants, modifier genes, genetic polymorphism, hormones, and lifestyle habits.) in women carrying BRCA1/2 variants.
3. To estimate the detection rates of occult cancer based on histopathological evaluations, using risk-reducing salpingo-oophorectomy (RRSO).
4. To examine the risk-reducing effect of RRSO on the development of ovarian, fallopian tube, and peritoneal cancers in women carrying BRCA1/2 variants, and compare with those not undergoing RRSO.
5. To identify clinicopathological features in women carrying BRCA1/2 variants who had undergone RRSO.
6. To identify the appropriate interval or degree of surveillance.

ELIGIBILITY:
Inclusion Criteria:

1. Women carrying BRCA1/2 variants (those with either BRCA1 or BRCA2 variants, or those carrying both variants) and women carrying a variant of uncertain significance (VUS).
2. Women who have received sufficient genetic counseling at any medical institution, prior to enrollment to the study.
3. Women who provide consent should be 20 years of age or older.
4. Women who provide written consent.

Exclusion Criteria:

1. Women without ovarian or fallopian tube cancer at the time of informed consent.
2. Women previously diagnosed with ovarian, fallopian tube, or peritoneal cancer, and not excluding those with a personal history of breast cancer development.
3. Other individuals considered inappropriate for involvement in this study by the investigator.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: BRCA1 and/or BRCA2 variant carriers
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-11-08 (Actual); Primary Completion 2032-03-31 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of ovarian, fallopian tube, and peritoneal carcinoma | up to 15 years
  Occurrence of ovarian, fallopian tube, and peritoneal carcinoma is a duration from the date of enrollment to the date of first occurrence of ovarian, fallopian tube, and peritoneal carcinoma. If the subjects have undergone RRSO, the duration is defined from the date of enrollment to the date of RRSO conduct

SECONDARY OUTCOMES:
Development of ovarian, fallopian tube, and peritoneal cancers, and the detection rate of occult cancer, based on evaluations of histopathological samples taken post-RSSO. | up to 15 years
  Development of ovarian, fallopian tube, and peritoneal cancers, and the detection rate of occult cancer is a duration from the date of enrollment to the date of first occurrence of ovarian, fallopian tube, and peritoneal carcinoma. If the subjects have undergone RRSO, the duration is defined from the date of enrollment to the date of RRSO conduct. The occult cancer is defined as ovarian, fallopian tube, peritoneal, and uterine carcinomas (including serious tubal intraepithelial carcinoma, STIC), which is based on evaluations of histopathological samples taken post-RSSO.
Death from any cause | up to 15 years
  Death from any cause is a duration from the date of enrollment to the date of death from any cause. If the subjects have undergone RRSO, the duration is defined from the date of enrollment to the date of RRSO conduct.
Deaths from ovarian, fallopian tube, and peritoneal cancers. | up to 15 years
  Deaths from ovarian, fallopian tube, and peritoneal cancers is a duration from the date of enrollment to the date of death from these cancers. If the subjects have undergone RRSO, the term is defined from the date of enrollment to the date of RRSO undergone.
Establishing the detection rate of occult cancer based on histopathological evaluations of samples from RRSO. | up to 15 years
  The occult cancer is defined as ovarian, fallopian tube, peritoneal, and uterine carcinomas (including serious tubal intraepithelial carcinoma, STIC), which is based on evaluations of histopathological samples taken post-RSSO.
Development of ovarian, fallopian tube, and peritoneal cancers, including in the post-RRSO period. | up to 15 years
  Development of ovarian, fallopian tube, and peritoneal cancers, including in the post-RRSO period is a duration from the date of enrollment to the date of first occurrence of ovarian, fallopian tube, and peritoneal cancer, including in the post-RRSO period.
Death from any cause, including post-RRSO period. | up to 15 years
  Death from any cause, including post-RRSO period is a duration from the date of enrollment to the date of death from any cause, including in the post-RRSO period.

CONTACTS AND LOCATIONS:
Overall Officials: Akira Hirasawa, M.D., Ph.D., Study Chair — Okayama University
Locations (1):
- Okayama University, Okayama, Japan